CLINICAL TRIAL: NCT00931021
Title: Smoking Cessation Treatment for Head and Neck Cancer Patients
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0903004910
Record Dates: First submitted 2009-06-29; First posted 2009-07-02 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Varenicline (Chantix) (Active Comparator)
  Interventions: Drug: Varenicline (Chantix)
- Nicotine Patch (Active Comparator)
  Interventions: Drug: Nicotine Patch

INTERVENTIONS:
Drug: Varenicline (Chantix) — 2 mg
  Other Names: Chanitx
  Arms: Varenicline (Chantix)
Drug: Nicotine Patch — 21 mg
  Arms: Nicotine Patch

SUMMARY:
This is a pilot research study examining the use of varenicline (Chantix) and the nicotine patch. The study is designed to find out whether one of these medications is more effective for smoking cessation with head and neck cancer patients. The study has three parts: 1) two intake sessions; 2) an 8-week treatment phase, and 3) a 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* smoking 10 or more cigarettes per day
* diagnosed with and completed an initial course of treatment for any type of head and neck cancer
* life expectancy of 12 months or more

Exclusion Criteria:

* history of allergic reactions to adhesives
* unstable psychiatric/medical conditions such as suicidal ideation, acute psychosis, severe alcohol dependence, or dementia
* females of childbearing potential who are pregnant, nursing, or not practicing effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To develop an effect size estimate for smoking cessation defined as continuous abstinence over the last 4 weeks of treatment for 2 mg varenicline compared to nicotine patch. | Eight weeks

SECONDARY OUTCOMES:
To examine tolerability of 2 mg varenicline and the 21 mg nicotine patch in smokers who have been diagnosed with head and neck cancer. | Eight weeks
To examine the effects of smoking cessation, varenicline and nicotine patch on markers of inflammation. | Eight weeks
To examine the effect of varenicline and nicotine patch on alcohol consumption. | Eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Toll, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States